CLINICAL TRIAL: NCT00876707
Title: Phase 1 Study of Ocular Aberrations and Visual Performance of Eyes Implanted With Three Multifocal Intra-ocular Lenses
Brief Title: Wavefront Analyzes and Visual Performance of Three Multifocal Intra-ocular Lenses
Acronym: IOL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Marcony Rodrigues de Santhiago, University of São Paulo
Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0088/09
Record Dates: First submitted 2009-04-03; First posted 2009-04-07 (Estimated); Last update posted 2010-07-02 (Estimated); Status verified 2009-04

CONDITIONS: Cataract; Astigmatism
Keywords: wavefront; multifocal IOL; modulation transfer function; intraocular lenses; wavefront data; Visual performance
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Who Masked: Investigator

ARMS (3):
- Tecnis (Active Comparator)
  Interventions: Device: Tecnis implant
- ReSTOR (Active Comparator)
  Interventions: Device: ReSTOR implant
- ReZoom (Active Comparator)
  Interventions: Device: ReZoom implant

INTERVENTIONS:
Device: Tecnis implant — Implant of diffractive multifocal IOL Tecnis
  Arms: Tecnis
Device: ReSTOR implant — Implant of multifocal IOL ReSTOR
  Arms: ReSTOR
Device: ReZoom implant — Implant of multifocal IOL ReZoom
  Arms: ReZoom

SUMMARY:
The purpose of this study is to determine if differences in the design of multifocal intra-ocular lenses would mean different values of higher-order aberrations and different performance in objective parameters such as modulation transfer function.

ELIGIBILITY:
Inclusion Criteria:

* Patients with bilateral visually significant cataract with corneal astigmatism lower than 1.0D

Exclusion Criteria:

* Any ocular diseases, such as:

  * corneal opacities or irregularity
  * dry eye
  * amblyopia
  * anisometropia
  * glaucoma
  * retinal abnormality
* Surgical complications
* IOL tilt
* IOL decentration greater than 0.4 mm (estimated by retroillumination)
* Incomplete follow-up

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
visual acuity, wavefront data and modulation transfer function | 30, 90 and 120 days after surgery

SECONDARY OUTCOMES:
contrast sensitivity | 90 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- University of São Paulo, São Paulo, São Paulo, Brazil